CLINICAL TRIAL: NCT00141401
Title: An Open-Label, Extension Safety and Efficacy Study of Pregabalin in Patients With Painful Diabetic Peripheral Neuropathy.
Brief Title: Safety and Efficacy of Pregabalin in Patients With Diabetic Peripheral Neuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-074
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate long-term efficacy and safety of pregabalin in patients with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for preceding double-blind study
* Must have received pregabalin or amitriptyline or placebo under double-blind conditions under double-blind conditions at least during first 3 weeks if double-blind treatment phase of preceding study.

Exclusion Criteria:

* Patients cannot be included if they experienced a serious adverse event while participating in preceding double-blind study, which was determined to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 1999-09; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer